CLINICAL TRIAL: NCT03027479
Title: Study of Differences in Skeletal Muscle Energy Metabolism Alterations in Women With Weight Loss and Ovarian and/or Endometrial Cancer Based on the Body Mass Index
Brief Title: Skeletal Muscle Energy Metabolism in Women With Weight Loss and Ovarian and/or Endometrial Cancer With Weight Loss
Acronym: METERMUS-IMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Inserm U1069 - Team Nutrition, Growth and Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PHAO16-LO/METERMUS-IMC; 2016-A01323-48 (Registry Identifier: IdRCB); 2016-R27 (Other: CPP)
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Weight Loss; Ovarian Carcinoma; Endometrial Carcinoma
Keywords: weight loss; ovarian cancer; endometrial cancer; energy metabolism; Body mass index; obesity; muscle energy
MeSH Terms: conditions — Weight Loss; Ovarian Neoplasms; Endometrial Neoplasms; Obesity | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): women with ovarian and/or endometrial cancer and weight loss will have muscle, adipose tissue, ovarian tumor and blood samples
  Interventions: Other: Samples
- Control group (Other): women scheduled for an intervention for benign ovarian/ endometrial disease and no weight loss will have muscle, adipose tissue and blood samples
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — Blood samples, muscle biopsy, adipose tissue samples and ovarian cancer tumor sample

SUMMARY:
the aim is to study skeletal muscle metabolism alterations métaboliques associated with weight loss in women with ovarian and/or endometrial cancer according to BMI.

ELIGIBILITY:
Case group selection criteria:

Inclusion Criteria:

* Women aged 18 years old and more
* Ovarian and/or endometrial cancer
* weight loss related to cancer (weight loss > 5% weight in one month or 10% in 6 months)
* Indication to therapeutic surgery
* Women affiliated to social security scheme
* Women who can understand French and able to sign Informed consent

Exclusion Criteria:

* Unbalanced Diabetes
* Chronic neuromuscular disorder
* Any severe uncontrolled medical condition

Control group selection criteria:

Inclusion Criteria:

* Women aged 18 years and more
* Surgery Indication for a benign endometrial and/ or ovarian disease
* Patient affiliated to social security scheme
* Women who can understand French and able to sign Informed consent

Exclusion Criteria:

* Unbalanced Diabetes
* Chronic neuromuscular disorder
* Any severe uncontrolled medical condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Measurement of muscle mitochondrial bioenergetics according to BMI | muscle biopsy realized during surgery
  Measurement of muscle mitochondrial bioenergetics by high resolution oxygraphy

SECONDARY OUTCOMES:
on muscle biopsy | muscle biopsy realized during surgery
  * Quantification of lipids on electron microscope
  * Type of muscular fibers
  * Analyze of gene expression and proteins involved in 1/ Mitochondrial metabolism 2/ lipid metabolism and 3/ muscular proteolysis by RTqPCR with SyBR Green and Western Blot
on white adipose tissue | adipose tissue samples taken during surgery
  adipose tissue composition (fatty acids quantification, sterols, steroids)
  * RT-qPCR quantification of molecules involved in lipid metabolism (synthesis, transport) and in inflammation (immune profile and cytokines)
  * RTqPCR analysis, western blot and immunohistochemical expression of markers of transformation into brown adipose tissue
  * in specific milieu, in vitro experimentation on skeletal muscular cells
on ovarian cancer tumor samples | ovarian tumor biopsies realized during surgery
  * lipid composition (fatty acids quantification, sterols, steroids)
  * RT-qPCR quantification of molecules involved in lipid metabolism (synthesis, transport) and in inflammation (immune profil and cytokines)
  * culture of tumour cells to evaluate resistance to chemotherapy (platinum)
on computerized tomography | 1 day of abdominal CT scan imaging procedure performed at diagnosis
  assessment of body composition (fat and muscle compartments)

CONTACTS AND LOCATIONS:
Overall Officials: Lobna OULDAMER, MD, PhD, Principal Investigator — University Teaching Hospital of Tours
Locations (1):
- Gynecology Department, University Teaching Hospital, Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salaun H, Poisson M, Dolly A, Arbion F, Servais S, Dumas JF, Goupille C, Ouldamer L. Total Polyunsaturated Fatty Acid Level in Abdominal Adipose Tissue as an Independent Predictor of Recurrence-Free Survival in Women with Ovarian Cancer. Int J Mol Sci. 2023 Jan 16;24(2):1768. doi: 10.3390/ijms24021768. PMID 36675280